CLINICAL TRIAL: NCT01678742
Title: Effects of Jeju Red Horsehead Fish-based, High Protein Diet on Satiety and Incretin Hormones in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeju National University Hospital (Other)
Responsible Party: Principal Investigator, Gwanpyo Koh, Associate professor, Jeju National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-06-007-002; C0038345 (Other Grant/Funding Number: The Small & Medium Business Administration)
Record Dates: First submitted 2012-08-25; First posted 2012-09-05 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: Diet; Incretins; Gastrointestinal Hormones; Fish Proteins
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-protein diet (Experimental)
  Interventions: Dietary Supplement: High-protein diet
- Standard diet (Active Comparator)
  Interventions: Dietary Supplement: Standard diet

INTERVENTIONS:
Dietary Supplement: High-protein diet — The high-protein diet is made up of 50% carbohydrate, 40% of protein and 10% of fat, providing 480 kcal.
  A protein part of the high-protein diet is mostly composed of a grilled Jeju red horsehead fish, a special product of Jeju island in Korea.
  Other Names: A Jeju red horsehead fish-based meal
  Arms: High-protein diet
Dietary Supplement: Standard diet — The standard diet is made up of 60% carbohydrate, 20% of protein and 20% of fat, providing 480 kcal.
  Other Names: A mixed meal
  Arms: Standard diet

SUMMARY:
The aim of our study is to investigate the effects of high-protein diet on satiety and incretin hormones in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Subjects signed a written informed consent form

Exclusion Criteria:

* Liver cirrhosis
* Chronic renal disease (serum creatinine > 2mg/dL)
* Severe congestive heart failure
* Significant infectious or inflammatory diseases
* intractable malignant neoplasm
* Pregnancy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Difference in the incremental area under the curve (iAUC) for peptide YY (PYY) after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.

SECONDARY OUTCOMES:
Difference in the iAUC for cholecystokinin (CCK) after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.
Difference in the iAUC for ghrelin after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.
Difference in the iAUC for glucagon-like peptide 1 (GLP-1) after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.
Difference in the iAUC for glucose-dependent insulinotropic polypeptide (GIP) after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.

OTHER OUTCOMES:
Difference in the iAUC for glucose after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.
Difference in the iAUC for insulin after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.
Difference in the iAUC for C-peptide after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.
Difference in the iAUC for glucagon after food ingestion between high-protein and standard diet groups | 3 hours
  Blood samples were drawn before the test meal (time 0) and at 30, 60, 90, 120, and 180 min after the test meal commenced.

CONTACTS AND LOCATIONS:
Overall Officials: Gwanpyo Koh, Professor, Principal Investigator — Jeju National University Hospital
Locations (1):
- Jeju National University Hospital, Jeju City, South Korea